CLINICAL TRIAL: NCT02984553
Title: The Use of Lactate Thresholds to Individualize Accelerometer Cut-points and Objectively Assess Physical Activity Levels in Postmenopausal Women
Brief Title: Objective Physical Activity Assesment in Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro de Estudios, Investigación y Medicina del Deporte (Other Government)
Collaborators: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Erreka Gil Rey, Principal Investigator, University of the Basque Country (UPV/EHU)
Other Study IDs: ACC-01
Record Dates: First submitted 2016-11-24; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Primary Prevention
Keywords: accelerometry; aerobic fitness; metabolic thresholds; moderate to vigorous physical activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to accurately assess weekly physical activity levels of postmenopausal women using lactate thresholds to individualize the accelerometer cut-points.

DETAILED DESCRIPTION:
This observational study aims to accurately assess weekly physical activity levels of postmenopausal women using lactate thresholds to individualize the accelerometer cut-points.

Postmenopausal women will be recruited from local advertisements in public health centers. Each woman will perfom on different days a progressive discontinuous submaximal walking-running test and several constant speed tests wearing an accelerometer to identify the individual lactate threshold (LT), the maximal lactate steady state (MLSS) and the corresponding accelerometer activity counts/min (cpm). Participants then will wear an actigraph accelerometer (wGT3X-BT) for seven days.

Linear regression equations will be developed for each participant to determine accelerometer activity counts for each intensity level: 1) sedentary behaviour (<200 cpm), 2) light intensity (200 cpm to activity counts at LT), 3) moderate intensity (activity counts between LT and MLSS) and 4) vigorous intensity (activity counts >MLSS). Physical activity levels will be measured using both, individualized approach and Sasaki, Jonh and Freedson´s (2011) absolute cut-points obtained through walking and running activities eliciting 3-6 MET intensities (2689-6166 cpm), considering it a "moderate" effort.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 70 years
* Surgical or natural menopause (no menstrual periods during at least the last 6 months)

Exclusion Criteria:

* Body mass index less than 39kg/m2 (obesity class III)
* Osteoporosis
* Presence of low-trauma fractures or severe arthrosis at hip, knees or feet
* Functional limitation to walk fast or altered gait patters and instability
* Presence of any chronic disesase that would impair the cardiovascular (e.g. myocardial infarction, stroke, chronic heart failure), musculoskeletal (osteoporosis, low-trauma fractures) and respiratory systems (COPD) or any disease or medication known to affect bone metabolism (glucocorticoids)

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Time spent in moderate-to-vigorous physical activities | 1 week
  The time spent in moderate-to-vigorous physical activities during a week (The participants have to wear an accelerometer attatched at the hip on an elastic belt for a period of 7 days)

SECONDARY OUTCOMES:
accelerometer intensity cut-points | an average of 1 month
  accelerometer activity counts corresponding to each woman´s lactate thresholds will determine each intensity level (These thresholds are determined on the walking-running tests performed on different days with a minimum of one week in between. These tests are independent, they are performed at constant speed during 20min to determine the highest speed at which the lactate concentration remains in a steady state between the minute 10 and 20 of the test)
Number of vertical acceleration peaks during the day | 1 week
  raw acceleration data will be measured to describe daily exposure to potentially osteogenic vertical impacts (The participants have to wear an accelerometer attatched at the hip on an elastic belt for a period of 7 days)
aerobic fitness | an average of 1 month
  determination of the speeds corresponding to the lactate thresolds during the walking-running test

OTHER OUTCOMES:
Maximum Strength | 1 day
  hand grip, leg and bench press maximum lifted weight (kg)
Heart rate variability | an average of 1 month
  the heart rate variability response during the walking-running tests and during the weekly physical activity assessment

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Gorostiaga, Medicine, Study Director — Centro de Estudios, Investigación y Medicina del Deporte
Locations (1):
- Centro de Estudios, Investigación y Medicina del Deporte, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: Yes
Codified IPD (personal data not shown, e.g. 321RR) will be shared with the Musculoskeletal Research Unit of the University of Bristol for the deep analysis of the 3th outcome

REFERENCES:
- [Background] Vainionpaa A, Korpelainen R, Vihriala E, Rinta-Paavola A, Leppaluoto J, Jamsa T. Intensity of exercise is associated with bone density change in premenopausal women. Osteoporos Int. 2006;17(3):455-63. doi: 10.1007/s00198-005-0005-x. Epub 2006 Jan 11. PMID 16404492
- [Background] Martyn-St James M, Carroll S. High-intensity resistance training and postmenopausal bone loss: a meta-analysis. Osteoporos Int. 2006;17(8):1225-40. doi: 10.1007/s00198-006-0083-4. Epub 2006 Jun 1. PMID 16823548
- [Background] Borer KT, Fogleman K, Gross M, La New JM, Dengel D. Walking intensity for postmenopausal bone mineral preservation and accrual. Bone. 2007 Oct;41(4):713-21. doi: 10.1016/j.bone.2007.06.009. Epub 2007 Jun 26. PMID 17686670
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Ozemek C, Cochran HL, Strath SJ, Byun W, Kaminsky LA. Estimating relative intensity using individualized accelerometer cutpoints: the importance of fitness level. BMC Med Res Methodol. 2013 Apr 1;13:53. doi: 10.1186/1471-2288-13-53. PMID 23547769
- [Background] Sasaki JE, John D, Freedson PS. Validation and comparison of ActiGraph activity monitors. J Sci Med Sport. 2011 Sep;14(5):411-6. doi: 10.1016/j.jsams.2011.04.003. Epub 2011 May 25. PMID 21616714
- [Background] Singh SJ, Morgan MD, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic airways obstruction. Thorax. 1992 Dec;47(12):1019-24. doi: 10.1136/thx.47.12.1019. PMID 1494764
- [Background] Miller NE, Strath SJ, Swartz AM, Cashin SE. Estimating absolute and relative physical activity intensity across age via accelerometry in adults. J Aging Phys Act. 2010 Apr;18(2):158-70. doi: 10.1123/japa.18.2.158. PMID 20440028
- [Background] Lopes VP, Magalhaes P, Bragada J, Vasques C. Actigraph calibration in obese/overweight and type 2 diabetes mellitus middle-aged to old adult patients. J Phys Act Health. 2009;6 Suppl 1:S133-40. doi: 10.1123/jpah.6.s1.s133. PMID 19998859
- [Background] Hannam K, Deere KC, Hartley A, Clark EM, Coulson J, Ireland A, Moss C, Edwards MH, Dennison E, Gaysin T, Cooper R, Wong A, McPhee JS, Cooper C, Kuh D, Tobias JH. A novel accelerometer-based method to describe day-to-day exposure to potentially osteogenic vertical impacts in older adults: findings from a multi-cohort study. Osteoporos Int. 2017 Mar;28(3):1001-1011. doi: 10.1007/s00198-016-3810-5. Epub 2016 Oct 31. PMID 27798733
- [Background] Beneke R. Methodological aspects of maximal lactate steady state-implications for performance testing. Eur J Appl Physiol. 2003 Mar;89(1):95-9. doi: 10.1007/s00421-002-0783-1. Epub 2003 Jan 21. PMID 12627312